CLINICAL TRIAL: NCT05331235
Title: Effect of Blood Transfusions on the Outcome of Low Birth Weight Preterm Infants
Brief Title: Blood Transfusions in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Douaa El Saied El Sherbiny, Lecturer of Pediatrics, Cairo university, Kasr El Aini Hospital
Other Study IDs: MS-49-2020
Record Dates: First submitted 2022-03-20; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Red Blood Cells; Preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross sectional study to assess the effect of blood transfusions on the outcome of preterm infants

DETAILED DESCRIPTION:
This is a cross sectional study carried on preterm infants who are staying in the hospital as "growers"; to gain weight. We will assess blood transfusion received by these preterm infants in details.

ELIGIBILITY:
Inclusion Criteria:

* Grower preterm infants

Exclusion Criteria:

* Severe illness, Hypovolemic shock, Hypoxia, Oxygen therapy, Surgical intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants admitted to the "grower ward", directly after birth or after transfer from NICU
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | immediately before and immediately after blood transfusion
  Heart rate per minute
Change in respiratory rate | immediately before and immediately after blood transfusion
  Respiratory rate per minute
Change in weight gain | within 4 days before and within 4 days after blood transfusion
  Average weight gain in grams/kg/day
Change in hemoglobin | immediately before and immediately after blood transfusion
  Hemoglobin in grams/dl
Change in hematocrit value | immediately before and immediately after blood transfusion
  Hematocrit value percentage

SECONDARY OUTCOMES:
Acute blood loss | in the previous 24 hours before blood transfusion
  Acute blood loss either spontaneous or iatrogenic during invasive procedures
Mechanical ventilation | in the previous 24 hours before blood transfusion
  Mechanical ventilation (MV) which may be one of two possibilities:
  1. Moderate or significant MV; Mean airway pressure (MAP) >8 cm H2O on conventional ventilator or >14 cm H2O on high frequency ventilator and FiO2 >0.4
  2. Minimal MV; MAP ≤8 cmH2O on conventional ventilator or ≤14 cm H2O on high frequency ventilator and FiO2 ≤ 0.4
Supplemental oxygen | in the previous 24 hours before blood transfusion
  Supplemental oxygen, not mechanically ventilated
Doubling of oxygen requirements | in the previous 2 days before blood transfusion
  Doubling of oxygen requirements for patients on supplemental oxygen
Tachycardia | in the previous 24 hours before blood transfusion
  ≥24 hours of tachycardia (Heart rate>180/minute)
Tachypnea | in the previous 24 hours before blood transfusion
  ≥24 hours of tachypnea (Respiratory rate>60/minute),
Poor weight gain | in the previous 4 days before blood transfusion
  ≤10 g/kg/day while the infant is receiving ≥120 kcal/kg/day
Metabolic acidosis | in the previous 24 hours before blood transfusion
  pH <7.2
Apnea and bradycardia | in the previous 24 hours before blood transfusion
  9 episodes or ≥2 episodes requiring bag and mask ventilation, while infant is receiving caffeine citrate
Length of stay in the NICU | from date of birth until the date of transfer to the "grower ward" or date of death from any cause, whichever came first, assessed up to 3 months.
  Length of stay in the NICU
Length of stay in the hospital | from date of birth until the date of discharge home or date of death from any cause, whichever came first, assessed up to 3 months.
  Length of stay in the hospital
Mortality | from the date of transfer to grower ward, assessed up to 3 months.
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Dahlia El Sebaie, MD, Study Director — Kasralainy hospital, Faculty of medicine, Cairo University

IPD SHARING:
Plan to Share IPD: Undecided